CLINICAL TRIAL: NCT06161610
Title: Randomized Clinical Trial of Efficiency and Safety of Recurrent High Grade Glioma Treated by Laser Interstitial Thermal Therapy
Brief Title: Recurrent High Grade Glioma Treated by LITT
Acronym: REGALITT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Dabiao Zhou, MD, MD, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REGALITT
Record Dates: First submitted 2023-11-21; First posted 2023-12-08 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Recurrent High Grade Glioma
Keywords: laser interstitial thermal therapy; Recurrent High Grade Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The progression will be assessed by third-party blinded investigators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LITT (Experimental): LITT+potential other treatment
  Interventions: Device: LITT
- Control (Active Comparator): Best medical management under guidelines
  Interventions: Other: Control

INTERVENTIONS:
Device: LITT — The patients in the intervention group will receive LITT, other treatments, including systematic therapy and radiology therapy, would be not restricted except the craniotomy of resection before tumor progression or emergency. The patient is supposed to receive LITT post-randomization within 7 days.
  Arms: LITT
Other: Control — The patients in the control group will receive the best medical management under guidelines except LITT before tumor progression. Craniotomy will not be restricted,
  Arms: Control

SUMMARY:
This clinical trial aims to investigate the efficiency and safety of laser interstitial thermal therapy (LITT) in recurrent high-grade glioma (rHGG) patients.

The main questions it aims to answer are:

* The LITT would increase the progression-free survival and overall survival of rHGG patients compared to other treatments.
* The LITT is safe and applicable to rHGG patients Participants will be randomized to the intervention group (LITT) or control group at a ratio of 2:1. The intervention group patients will receive LITT. The control group will be treated with any other treatment.

The primary outcome of this trial is progression-free survival. The estimated sample size is 135, 90 in the LITT group and 45 in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years old or above;
2. Patients with previous pathological diagnosis of 2021 World Health Organization Classification of Central Nervous System Tumors (WHO CNS5) grade 3 or 4 glioma and received standard treatment;
3. Meet any of the following:

   1. Meets the disease progression criteria in the Response Evaluation of Neuro-Oncology (RANO 2.0) criteria;
   2. At least one image other than T1 contrast indicates progression;
   3. Pathology shows progression or recurrence;
   4. Other progress determined by the Clinical Events Committee (CEC);
4. All tumor lesions are located supratentorial and the maximum cross-sectional short-axis length in the T1 contrast is ≤30 mm;
5. Karnofsky score (KPS) ≥ 60 and the patient can tolerate the intervention;
6. The subjects or their agent can understand the purpose of the trial, show sufficient compliance with the trial protocol, and sign the informed consent form.

Exclusion Criteria:

1. Patients may benefit from other treatments or may not benefit from this trial;
2. No more than three months since the patient underwent craniotomy;
3. MRI contrast cannot be performed;
4. Severe coagulation disorder;
5. Women who are pregnant, lactating, or planning to become pregnant within 6 months;
6. Participated in any other clinical trials of drugs or medical devices within 3 months;
7. Combined diseases that may interfere with treatment or prognosis assessment;
8. Refuse or unlikely to complete follow-up assessment;
9. Other circumstances in which the researcher deems it inappropriate to participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2027-09-19 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | estimate 6 months
  The progression was defined by RANO 2.0 criteria and assessed by the third-party clinical events committees which are blinded to the allocation.

SECONDARY OUTCOMES:
Lesion ablation rate | within 2 days Post LITT
  LITT group only, measured on enhanced MRI within 2 days post LITT
Lesion remaining volume | within 2 days Post LITT
  LITT group only, measured on enhanced MRI within 2 days post LITT
Overall survival | up to 2 years
Karnofsky Performance Status (KPS) shift | Day 30,Day 90, Day 180
  The difference between baseline KPS and follow-up KPS

OTHER OUTCOMES:
specific AE rate | through study completion, an average of 6 month
  Specific AE and complication including intracerebral hemorrhage, severe edema, newly seizure, local incision wound and all SAEs
bleeding volume | post LITT immmediatly
  LITT group only during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (9):
- China (9):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Wuhan, Hubei
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Peoples Hospital of Liaoning, Shenyang, Liaoning
  - Qilu Hospital, Jinan, Shandong
  - Huashan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No